CLINICAL TRIAL: NCT03096340
Title: A Phase 1 With Expansion Cohort, Open-Label, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of Intravenously Infused IT-141 in Subjects With Recurrent or Refractory Solid Tumors
Brief Title: Safety and Pharmacokinetic Study of IT-141 in Monotherapy in Patients With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated by sponsor.
Sponsor: Intezyne Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IT141-001
Record Dates: First submitted 2017-03-15; First posted 2017-03-30 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-01

CONDITIONS: Cancer; Neoplasms; Tumors; Refractory Solid Tumors; Recurrent Solid Tumors
Keywords: SN-38; irinotecan
MeSH Terms: conditions — Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IT-141 (Experimental)
  Interventions: Drug: IT-141

INTERVENTIONS:
Drug: IT-141 — Escalating doses administered in mg/m2, IV (in the vein) on days 1 and 15 of each 28 day cycle until progression or unacceptable toxicity develops.
  Other Names: IT-141, 7-ethyl-10-hydroxycamptothecin

SUMMARY:
IT141 is a novel nanoparticle formulation of SN-38, the active metabolite of irinotecan, and is intended to deliver more drug to the tumor with reduced toxicity on normal tissues. The study is designed to determine the maximum tolerated dose (MTD) of IT-141, and to investigate pharmacokinetic (PK) parameters and possible pharmacodynamics (PD) relationships. Patients will also be monitored for any response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older.
* Must be males or non-pregnant females who agree to comply with applicable contraceptive requirements of the protocol.
* Must have a histologically or cytologically confirmed, incurable malignancy, for which further standard treatment is not currently available.
* Must have measurable or evaluable disease during the dose escalation phase (measurable disease is preferred for the expanded cohort after MTD is reached).
* Must have an anticipated survival of at least 12 weeks.
* Must be fully informed regarding their illness and the investigational nature of the study protocol, and must sign an Institutional Review Board (IRB) approved Informed Consent Form (ICF).
* Must be ambulatory, with an Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1.
* Must have adequate organ function, as defined by the following:
* Hematologic: ANC 1.5 x 109/L, Hgb ≥ 9.0 g/dL and platelet count 100 x 109/L (platelet count > 75 x 109/L if documented evidence of bone marrow involvement).
* Hepatic: Total bilirubin 1.5 x ULN; transaminases ≤ 2.5 x ULN (may be up to 5 x ULN if clearly due to liver metastases); prothrombin time (PT) and partial thromboplastin time (PTT) < 2 x (ULN).
* Renal: Serum creatinine 1.5 x ULN or creatinine clearance 60 mL/min.
* Must be on stable doses of any drugs affecting hepatic drug metabolism or renal drug excretion (e.g. non-steroidal anti-inflammatory drugs, corticosteroids, barbiturates, diphenylhydantoin, narcotic analgesics, probenecid). Such drugs should not be initiated less than 30 days prior to Baseline/C1D1 or at any time during study participation. Whenever possible, narcotic analgesic doses should be stable within 30 days prior to study entry and during the first cycle of therapy.
* Must be recovered from any reversible side effects of prior therapy (e.g. no major surgery, no antineoplastic or experimental therapy, or no significant radiation therapy to hematopoietic sites within 4 weeks of Baseline/C1D1, and no nitrosoureas or nitrogen mustards within 6 weeks of Baseline/C1D1)
* Must understand and be able, willing, and likely to fully comply with study procedures and restrictions.

Exclusion Criteria:

* Current or recurrent disease that could affect the action or disposition of IT-141, or clinical or laboratory assessments.
* Subjects with UGT1A1*28 polymorphisms.
* Current or relevant previous history of serious, severe or unstable (acute or progressive) physical or psychiatric illness, including any medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that presents undue risk from the IP or procedures.
* Primary brain tumors or known brain metastasis unless clinically stable and on stable or reducing doses of steroids.
* Frequent vomiting.
* Recent history of unintentional weight loss > 10% of current body weight in the past 3 months.
* Ongoing radiation therapy, chemotherapy, or hormonal therapy. Point radiation to a site of bone pain will be allowed.
* Current (within 1 week of Screening) or regular use of any medication (including over-the-counter (OTC), herbal or homeopathic preparations) that could improve or worsen the cancer being studied, or could affect the action or disposition of IT-141, or its clinical or laboratory assessment; e.g. Coumadin therapy, due to high competitive protein binding. Subjects taking ANY supplemental IRON, i.e., therapeutic or as part of a multivitamin regimen, are excluded from this study, whether prescribed or self-medicated.
* Concomitant use of a UGT1A1 inhibitor, such as idinavir, atazanavir and sorafenib, throughout the study period.
* Known or suspected intolerance or hypersensitivity to IT-141 or any of the stated ingredients.
* History of alcohol or other substance abuse within the last year.
* History of use of another IP within the last 4 weeks prior to enrollment.
* Female subjects who are pregnant or lactating, including females with a positive pregnancy test at screening.
* Previous enrollment in this study, followed by withdrawal for any reason.
* Known HIV-positive subjects on combination anti-retroviral therapy due to the potential for PK interactions with the study agent.
* Evidence of ischemia or myocardial infarction within the past 6 months, or any significant abnormality on ECG.
* A QTc interval outside of normal. (Normal: < 450 msec for males and < 460 msec for females)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of IT-141 administered once every 2 weeks in patients with refractory solid tumors | 18 months

SECONDARY OUTCOMES:
Adverse event profiles according to the Common Toxicity Criteria for Adverse Events (CTCAE, ver. 4.03) | 18 months
Objective response rate based on RECIST | 18 months
Area under the plasma concentration versus time curve (AUC) of SN-38 and SN-38G | 18 months
Maximum plasma concentration (Cmax) of SN-38 and SN-38G | 18 months
Time to Cmax (Tmax) of SN-38 and SN-38G | 18 months
Elimination rate constant of SN-38 and SN-38G | 18 months
Terminal half-life (t1/2) of SN-38 and SN-38G | 18 months
Total plasma clearance (CL) of SN-38 and SN-38G | 18 months
Volume of distribution (Vz) of SN-38 and SN-38G | 18 months

OTHER OUTCOMES:
Overall Survival | 18 months
Progression-free Survival | 18 months
Time to progression | 18 months
Disease Control Rate | 2 years
MRI imaging for biodistribution of IT-141 | 18 months
Presence of cfDNA | 2 years
Presence of exosomes | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Minal Barve, MD, Principal Investigator — Mary Crowley Cancer Research Centers - Medical City; Kit Wong, MD, Principal Investigator — Seattle Cancer Care Alliance
Locations (2):
- United States (2):
  - Mary Crowley Cancer Research Centers - Medical City, Dallas, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bakewell SJ, Carie A, Costich TL, Sethuraman J, Semple JE, Sullivan B, Martinez GV, Dominguez-Viqueira W, Sill KN. Imaging the delivery of drug-loaded, iron-stabilized micelles. Nanomedicine. 2017 May;13(4):1353-1362. doi: 10.1016/j.nano.2017.01.009. Epub 2017 Jan 20. PMID 28115246